CLINICAL TRIAL: NCT01248312
Title: Estimation of the Incidence of Hypercapnea in Morbidly Obese Post-Surgical Patients Using the Sen Tec Transcutaneous PCO2 Monitor
Brief Title: Incidence of Hypercapnea in Morbidly Obese Post-Surgical Bariatric Patients Using the Sen Tec Transcutaneous PCO2 Monitor
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Roy Soto, MD, Principal Investigator, Corewell Health East
Other Study IDs: 2010-208
Record Dates: First submitted 2010-11-17; First posted 2010-11-25 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Bariatric Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- morbidly obese: BMI >45
  Interventions: Device: Sentec monitoring device; Device: sentec monitor
- thin patients: BMI <45
  Interventions: Device: Sentec monitoring device; Device: sentec monitor

INTERVENTIONS:
Device: Sentec monitoring device — Sentec monitor applied transcutaneously to forehead
Device: sentec monitor — transcutaneous monitoring
  Other Names: Sentec monitoring device

SUMMARY:
Hypercapnea is a condition where there is too much carbon dioxide (CO2) in the blood. Carbon dioxide is a gaseous product of the body's metabolism and is normally expelled through the lungs (breathed out). Hypoventilation (or respiratory depression) occurs when the ventilation is inadequate to perform needed gas exchange; therefore resulting in decreased levels of oxygen and increased levels of carbon dioxide in the blood. It can cause an increased concentration of carbon dioxide and respiratory acidosis. Obesity is a multi-system disorder, particularly involving the respiratory (lungs/breathing) and cardiovascular (heart/vessel) systems. Obesity increases the risks for surgical and anesthetic complications before, during and following surgery.

Bariatric (weight loss) surgery is becoming a common procedure among the morbidly obese (100 lbs or more above normal weight), with recent studies highlighting the long-term health implications of surgical weight reduction, to include a decreased risk of hypertension (high blood pressure) and diabetes (increased sugar in blood). Obese patients are at increased risk of sleep apnea (stop breathing while asleep) and hypoventilation even without surgery, and these risks increase following administration of medications typically given during and after major surgical procedures. Hypoventilation can lead to hypercapnea, sedation (sleepiness), and acidosis (blood imbalance), resulting in further respiratory compromise (breathing problems) and cardiac morbidity (heart problems) as well as the risks inherent in re-intubating (needing to have a breathing tube place down into the lungs) the obese.Monitoring for hypoventilation can be difficult. Quantitative capnography (measuring carbon dioxide) is only appropriate for intubated patients (on a ventilator - breathing tube), and pulse oximetry (clip on finger that measures oxygen levels) does not adequately detect hypoventilation in patients receiving supplemental (additional) oxygen. Serial arterial blood gas (blood taken from an artery to measure oxygen level in blood) measurement is expensive, time-consuming, and painful. Continuous respiratory rate monitoring is possible, and has been considered the gold standard of apnea detection (seeing stopped breathing), yet is seldom used. As a result of these limitations, there is currently no simple, cost-effective, and reliable means of detecting hypoventilation in this patient population either in the recovery room or inpatient unit. Transcutaneous (across the skin) pCO2 (t-pCO2) monitoring has been validated as a reliable and reproducible means of measuring pCO2 in newborn babies, and recently has also been used in adults, primarily in the ICU (intensive care unit) setting. When compared to standard end-tidal CO2 measurement, t-pCO2 correlates better with pCO2 in the intraoperative period in both thin and obese patients. SenTec, is the manufacturer of a device used to measure t-pCO2 for this project. This study is designed to detect the incidence of hypercapnea in morbidly obese post-surgical bariatric patients in the postoperative period using the SenTec t-pCO2 monitor.

Objective:To determine the incidence of hypoventilation and hypercapnea as measured by transcutaneous pCO2 monitoring in post-surgical bariatric patients as compared to thin controls.

ELIGIBILITY:
Inclusion Criteria:

* Consenting male or female adults aged 18-65, scheduled to undergo elective laparoscopic gastric bypass (morbidly obese) or patients scheduled to undergo an abdominal procedure (thin) which will similarly require an overnight admission to Beaumont/Royal Oak Hospital
* Women must be nonpregnant and nonlactating, postmenopausal or surgically sterile. Women of childbearing age must have a negative pregnancy test (performed per standard hospital protocol

Exclusion Criteria:

* History of COPD (lung/breathing disease)
* Home O2 (oxygen) dependence (home CPAP use is acceptable)
* Pregnancy/nursing
* Scheduled to receive epidural pain management.(Epidural pain management is the continuous infusion of medication(s) into the space surrounding the spinal cord called the epidural space.)
* Participation in another clinical trial within the past 30days
* Skin condition that would interfere with the application of the forehead sensor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 morbidly obese post surgical laparoscopic bariatric patients and 10 thin subjects undergoing laparoscopic procedures
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of hypoventilation and hypercapnea as measured by transcutaneous pCO2 monitoring in post surgical bariatric patients as compared to thin controls. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Roy Soto, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States